CLINICAL TRIAL: NCT02480699
Title: Intra Individual Evaluation of Uremic Toxin Levels in Hemodialysed Patients
Acronym: EVITUPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-10; 2015-A00319-40 (Registry Identifier: ANSM); RCAPHM15_0083 (Other: APHM)
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemodialysed patients (Experimental)
  Interventions: Biological: Recurring blood sample; Other: dietary survey

INTERVENTIONS:
Biological: Recurring blood sample
Other: dietary survey — A dietary survey will be performed in all patients and every 3 months (4 surveys about 1 year). This survey will be given to the patient filled for 7 consecutive days. He must record during these 7 days, all of his food intake in quality and quantity. During a dialysis session this questionnaire will be taken with the patient by a dietician to better define the food intake. This surveys requires good patient compliance as well as his involvement that his collection is well within its food intake.

SUMMARY:
Chronic kidney disease (CKD) is characterized by a irreversible decrease of kidney functions. It is characterized by accumulation of solutes called uremic toxins. Uremic toxins levels are implicated in cardiovascular complications associated with CKD. Several protein-bound toxins have been implicated in the increased cardiovascular risk such as indoxyl sulfate (IS), p cresol sulfate (pCS) and more recently the indole acetic acid (IAA). All clinical studies are performed with a single measurement at baseline assuming that the toxin levels are stable over time. The variability of uremic toxins level is not known. Furthermore, little is known concerning determinants of serum toxins level.

DETAILED DESCRIPTION:
Colonic absorption play a major role in IS (indoxyl sulfate) and pCS level. IS and pCS level are significantly reduced in patient with colectomy. To validate the measurement of uremic toxins level in serum as biomarkers for cardiovascular risk, we need to know about intra-individual variability over time and the impact of diet or digestive disorders on uremic toxin serum level. We propose a prospective study evaluating the intra-individual variability in 3 uremic toxins serum levels the SI, the pCS and IAA.

The main objective is to study the kinetics of three serum uremic toxins: the indoxyl sulfate, p cresyl sulfate and indole acetic acid (and thus determine the intra-individual variability) in a population of chronic hemodialysis patients during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Major subjects of both sexes aged 18 and over
* Topics affiliates or beneficiaries of a social security scheme
* Haemodialysis patients whatever the etiology of renal failure for more than 3 months
* Patients not under antibiotic
* Agreeing to participate in the study and who signed a consent
* Patient able to understand a written questionnaire

Exclusion Criteria:

* Pregnant or lactating women
* Detainees
* Adults under legal protection or unable to consent
* Patient's refusal to sign the informed consent for participation
* Possibility of recovery of renal function (eg scleroderma)
* Patients carrying a replicating viral infection (HCV, HIV).
* Taking antibiotics in the previous month by 1 sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-06-20 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Composite measure of uremic toxins serum levels the SI, the pCS and IAA. | 15 months
  blood collection

SECONDARY OUTCOMES:
dietary survey | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique H^^opitaux de Marseille, Marseille, France